CLINICAL TRIAL: NCT01134380
Title: Genotyping Infarct Patients to Adjust and Normalize Thienopyridine Treatment
Acronym: GIANT
Status: Completed | Type: Observational
Sponsor: Biotronik France (Industry)
Collaborators: European Cardiovascular Research Center (Network); Allies in Cardiovascular Trials Initiatives and Organized (Other)
Responsible Party: Virginie COLIN, Biotronik France
Other Study IDs: GIANT200905-04
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Genetic Resistance to Clopidogrel; Compliance to Thienopyridine Treatment
Keywords: Percutaneous coronary intervention; Acute coronary syndrome; Dual antiplatelet therapy; clopidogrel/prasugrel; genotyping; stent; compliance
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA Samples from saliva to observe CYP2C19 genetic variants
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- [*1] Genotype - Good responders to Clopidogrel: This group of patients is defined thanks to the DNA extracted from their saliva: [*1] genotype patients are good responders to clopidogrel
- [*2] genotype with adapted thienopyridine treatment: This group of patients is defined thanks to the DNA extracted from their saliva: [*2] genotype patients are bad responders to clopidogrel and their thienopyridine treatment has been adapted

SUMMARY:
The objective of GIANT Study is to evaluate the clinical impact of genetic resistance to thienopyridine profile determination (CYP2C19 gene) and the clinical impact of compliance to an adjusted thienopyridine treatment on STEMI patients treated by primary PCI within the 24 hours following the first chest pain.

DETAILED DESCRIPTION:
All the STEMI patients treated by primary PCI (with stent implantation) within the 24 hours following the first chest pain can be included in the GIANT study. After the PCI, they'll receive DAT (Aspirin + Clopidogrel/Prasugrel).

Patients will then be genotyped to determine if they carry one of the CYP2C19 gene variants making them resistant or hyper responder to clopidogrel. The genetic profile of the patients will be communicated to the physician who took care of them so that he can (or not) adjust the thienopyridine treatment (increase of the clopidogrel dosage, switch to prasugrel or switch to clopidogrel). A treatment will be prescribed for 12 months as according to the European guidelines.

One year after the PCI, the patients will have to be available for a follow up visit. They'll be submitted to a VERIFY NOW P2Y12 protocol to determine whether they were compliant to their thienopyridine treatment. A clinical follow up will be also performed to evaluate the cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patient treated within the first 24 hours with primary PCI (with stent implantation)
* Age superior or equal to 18 years old
* Informed consent signed
* Patient volunteer to be submitted to the 1 year visit follow up and to the clinical exams during this visit
* Patient benefiting from French social health system

Exclusion Criteria:

* NONSTEMI patient with high troponin
* STEMI patient treated after the first 24 hours
* Stable / unstable angina or silent ischemia
* Cardiogenic shock
* Oral anticoagulation (Vitamin K Antagonists)
* Contraindication for PCI
* Age inferior to 18 years old
* Life expectancy inferior to 1 year
* Participation in another clinical trial
* No signed informed consent
* Patient not available for the 1 year visit follow up
* Pregnant women
* Known allergy to media contrast that can not be controlled by an adapted treatment
* Known allergy to cobalt chromium alloy
* Left ventricular ejection fraction lower than 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: STEMI patients treated within the first 24 hours following the first chest pain by Primary PCI (with stent implantation)
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
statistical difference in Death, MI and stent thrombosis between genetically resistant patients (*2 genotype) with adapted treatment and non resistant patients (*1 genotype) | 12 months

SECONDARY OUTCOMES:
Difference in MACCE between responder + compliant patients vs responders + non compliant patients vs non responder patients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chevalier, Principal Investigator — Hopital Privé Jacques Cartier; Gilles Montalescot, Principal Investigator — Assistance Publique Hopitaux de Paris; Loïc Belle, Principal Investigator — Centre Hospitalier de la région Annecienne
Locations (12):
- France (12):
  - Centre Hospitalier de la Région Annecienne, Annecy
  - Hôpital Albert Schweitzer, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier d'Haguenau, Haguenau
  - Centre Hospitalier Saint Joseph et Saint Luc, Lyon
  - Hôpital Privé Jacques Cartier, Massy
  - Hôpital Bon Secours, Metz
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire Caremeau, Nîmes
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Centre Hospitalier Rene Dubos, Pontoise
  - CHI de Villeneuve, Villeneuve-Saint-Georges

REFERENCES:
- [Derived] Hulot JS, Chevalier B, Belle L, Cayla G, Khalife K, Funck F, Berthier R, Piot C, Tafflet M, Montalescot G; GIANT Investigators. Routine CYP2C19 Genotyping to Adjust Thienopyridine Treatment After Primary PCI for STEMI: Results of the GIANT Study. JACC Cardiovasc Interv. 2020 Mar 9;13(5):621-630. doi: 10.1016/j.jcin.2020.01.219. PMID 32139220